CLINICAL TRIAL: NCT07055360
Title: A Trauma-Informed Intervention for Sexual Minority Men Recently Diagnosed With HIV
Brief Title: A Trauma-Informed Intervention for the Newly HIV-Diagnosed
Acronym: RISE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34MH132561 (NIH); 1R34MH132561-01 (NIH)
Record Dates: First submitted 2025-04-07; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Stress; HIV Care Loss to Followup; HIV Treatment Cascade
Keywords: resilience; trauma; intervention; mental health; HIV; HIV care; newly-diagnosed; mHealth; eHealth; stress
MeSH Terms: conditions — Wounds and Injuries; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resilience-Based Intervention for Stress Reduction and HIV-Related Efficacy (RISE) (Experimental): Resilience-Based Intervention for Stress Reduction and HIV-Related Efficacy (RISE). RISE is based on Cognitive-Behavior Therapy (CBT) and the Information-Motivation-Behavioral Skills (IMB) Model. RISE will consist of six, weekly sessions, followed by a booster session in week 8, including resilience-building and health-promoting activities of RISE. Sessions will emphasize the participants' strengths, including positive thoughts, beliefs, and behaviors that work for the client and existing assets and supports in the participant's life. Tailored, health-promotion text messages will be sent weekly after each session.
  Interventions: Behavioral: Resilience-Based Intervention for Stress Reduction and HIV-Related Efficacy (RISE)
- Waitlist Control: Text messaging-reminder comparison condition (Active Comparator): This control condition will involve reminder text messages for adherence to HIV treatment and engaging in HIV care. This is a waitlist control condition, as participants in this condition will ultimately receive the intervention.
  Interventions: Behavioral: Waitlist control: Text messaging-reminder comparison condition

INTERVENTIONS:
Behavioral: Resilience-Based Intervention for Stress Reduction and HIV-Related Efficacy (RISE) — RISE is based on Cognitive-Behavior Therapy (CBT) and the Information-Motivation-Behavioral Skills (IMB) Model. RISE will consist of six, weekly sessions, followed by a booster session in week 8, including resilience-building and health-promoting activities of RISE. Sessions will emphasize the participants' strengths, including positive thoughts, beliefs, and behaviors that work for the client and existing assets and supports in the participant's life. Tailored, health-promotion text messages will be sent weekly after each session.
  Arms: Resilience-Based Intervention for Stress Reduction and HIV-Related Efficacy (RISE)
Behavioral: Waitlist control: Text messaging-reminder comparison condition — This control condition will involve reminder text messages for adherence to HIV treatment and engaging in HIV care. As this condition is a waitlist control, participants in this condition will ultimately receive the RISE intervention.
  Arms: Waitlist Control: Text messaging-reminder comparison condition

SUMMARY:
The current approach to HIV prevention emphasizes: (1) achieving viral suppression among HIV+ people in order to reduce HIV transmissibility, particularly for disproportionately affected groups such as Black sexual minority men (BSMM), by increasing retention in HIV care, and (2) addressing comorbidities and complications, which include mental health concerns such as trauma symptomology and severe acute stress reactivity. Despite the disproportionate impact of both HIV and traumatic stress on BSMM and the adverse effects of stress on engagement in HIV care, BSMM remain grossly underserved with respect to mental health. To address these gaps, the proposed study will develop an intervention that will: (1) provide a brief, resilience-oriented, trauma-informed intervention that combines online sessions and highly tailored text-messaging to reduce participant burden and motivate clients between sessions, (2) provide preliminary treatment for HIV+ BSMM's unaddressed mental health needs, and (3) be embedded early in the HIV continuum of care immediately after diagnosis to facilitate linkage to and retention in HIV care.

DETAILED DESCRIPTION:
Compared to the general population in the United States, people living with HIV (PLWH) show high rates of trauma- and stress-related disorders and severe acute stress reactivity to events that are, diagnostically, not considered traumatic. Trauma is highly correlated with depression, a robust predictor of antiretroviral treatment (ART) non-adherence. Additionally, reporting a high number of recent stressful events is associated with ART non-adherence. Despite Black sexual minority men (BSMM), particularly those under age 40, being disproportionately affect by HIV and trauma and less likely to be linked to HIV care after diagnosis, BSMM remain grossly underserved with respect to mental health. Further, although interventions exist that address trauma for PWLH, few HIV-related interventions emphasize the traumatic stress cycle and acute stress reactivity immediately following an HIV diagnosis. To address the need for early mental health intervention immediately after HIV diagnosis, in general, as well as the under-addressed mental-health needs of HIV+ BSMM (+BSMM), in particular, the investigators will develop and pilot-test a resilience-focused, trauma-informed intervention called, Resilience- Based Intervention for Stress Reduction and HIV-Related Efficacy (RISE). RISE will be based on approaches and techniques of Cognitive-Behavior Therapy (CBT) and the framework of Resilience Theory. It will address trauma- and stress-related symptomology and acute stress reactivity within three months of an HIV diagnosis to facilitate linkage to HIV care. The brief RISE will include six online sessions, a booster session, and text messaging. Innovative commercial marketing techniques will be used to develop highly targeted messages to supplement the CBT- and resilience-based approach of RISE. First, Aim 1 will involve formative research to assess +BSSM's needs, preferences, and perceptions regarding mental health and engagement in HIV care via in-depth interviews with +BSMM and service providers. Next, Aim 2 will include development of the RISE intervention manual and digital health infrastructure. Tailored text messages and health-promotion materials will be developed via in-depth interview-derived quantitative surveys with 50 +BSMM. The Aim will also include an iterative process of intervention development, including focus groups with +BSMM and service providers, respectively, and intervention theatre tests with 6 +BSMM. Finally, Aim 3 will consist of a randomized, controlled pilot trial for feasibility (e.g., recruitment and enrollment rates, fidelity), acceptability (i.e., feedback interview, satisfaction questionnaire), and preliminary efficacy (i.e., increased HIV care engagement, including attending an HIV care appointment, antiretroviral treatment ART initiation, and ART adherence primary outcome; reduced trauma symptoms, including intrusive experiences, avoidance, and hyperarousal secondary outcome) with 40 +BSMM diagnosed within the past three months. Participants will be assessed at baseline, post-intervention, and 6- and 9-month follow-ups post-baseline. The investigators will develop and maintain a community advisory board for consultation throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HIV within the past 3 months
* Self-identification as Black or African American
* Aged 18-39 years
* Elevated traumatic stress as indicated by scores above clinical cutoffs on either of the following subscales of the Impact of Event Scale--Revised: Intrusion (score of 5 or greater) and Avoidance (score of 7 or greater)
* Owning a phone with short-message service or messaging
* Access to a device with a screen, a web browser, and adequate internet speed for videoconferencing (e.g., smartphone, computer).

Exclusion Criteria:

* Demonstrating cognitive impairment or acute psychosis
* Reporting unvailability to participate in the Baseline Assessment, the RISE intervention, and 3-, 6, and 9-Month Follow-Up Assessments

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-09-12 (Estimated)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire-8 | Throughout study completion: 3-, 6- and 9-Month Follow-Up Post-Baseline
  Acceptability, specifically participant satisfaction. Values: Range from 8 to 32. Scoring: Higher scores indicate greater percentage of HIV medication dosages taken over the past 30 days.

SECONDARY OUTCOMES:
Question (Yes/No; Attended HIV care appointment in past 3 months): "Have [the participant] attended an HIV care appointment with a HIV care, primary care, or similarly care provider in the past 3 months?" | Throughout study completion: Baseline and 3-, 6- and 9-Month Follow-Up Post-Baseline
  Response options: Yes or No
Question (Yes/No; Initiated antiretroviral treatment): "Have [the participant] begun taking medication prescribed to treat HIV?" | Throughout study completion: Baseline and 3-, 6- and 9-Month Follow-Up Post-Baseline
  Response options: Yes or No
Question (Yes/No; Have future appointment scheduled): "Do [the participant] have a future HIV care appointment scheduled?" | Throughout study completion: Baseline and 3-, 6- and 9-Month Follow-Up
  Response options: Yes or No
Visual Analog Scale | Throughout study completion: Baseline and 3-, 6- and 9-Month Follow-Up Post-Baseline
  Antiretroviral treatment adherence for HIV (percentage). Values: Range from 0% to 100%. Scoring: Higher scores indicate greater percentage of HIV medication dosages taken over the past 30 days.
Berlin Social Support Scale | Throughout study completion: Baseline and 3-, 6- and 9-Month Follow-Up Post-Baseline
  Berlin Social Support Scales. Values: Range from 52 (minimum) to 208 (maximum). Scoring: Higher scores indicate greater social support (e.g., greater perceived support, greater desire for support, greater receipt of support, etc.), although some items need to be reverse coded.
Impact of Event Scale - Revised | Throughout study completion: Baseline and 3-, 6- and 9-Month Follow-Up Post-Baseline
  Traumatic stress symptomology, specifically avoidance and intrusion. 8 items ranging from 0 (minimum) to 32 (maximum) for avoidance and intrusionm respectively.
Center for Epidemiologic Studies - Depression Scale | Throughout study completion: Baseline and 3-, 6- and 9-Month Follow-Up Post-Baseline
  Depressive symptomology. Values: 20 items, range from 0 (minimum) to 60 (maximum) Scoring: Greater scores = more severe depression during the past week; 4 items (4, 8, 12, 16) need to be reverse coded
Beck Depression Inventory-II | Throughout study completion: Baseline and 3-, 6- and 9-Month Follow-Up Post-Baseline
  Depressive symptomology. Values: 21 items, range from 0 (minimum) to 63 (maximum). Scoring: Greater scores = greater depressive symptom severity.
Coping Self-Efficacy Scale | Throughout study completion: Baseline and 3-, 6- and 9-Month Follow-Up Post-Baseline
  Participants' belief in ability to cope. Values: 26 items, range from 0 (minimum) to 260 (maximum). Scoring: Greater scores = greater coping self-efficacy.
Illness Intrusiveness Ratings Scale | Throughout study completion: Baseline and 3-, 6- and 9-Month Follow-Up Post-Baseline
  Extent to which the illness reduces or intrudes upon quality of life. Values: 13 items, range from 13 (minimum) to 91 (maximum). Scoring: Greater scores = greater illness intrusiveness.
HIV Treatment Adherence Self-Efficacy Scale | Throughout study completion: Baseline and 3-, 6- and 9-Month Follow-Up Post-Baseline
  Participants' confidence in ability to adhere to antiretroviral treatment for HIV.
  Values: 12 items, range from 12 (minimum) to 120 (maximum). Scoring: Greater average scores = greater self-efficacy for treatment adherence in the past month.
Demographics | Baseline
  Participants enter or select demographic characteristics with which they identify, such as age, ethnicity, years of formal education, and annual household income.
Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) | Baseline
  Substance use severity based on the use of specific substances (i.e., alcohol, cigarette/nicotine smoking, and other substance, including illicit substances) endorsed by the participant.
  Values: For each drug, participants respond yes or no to any lifetime use. Subsequently, for each drug, participants complete six items with scores ranging from 0 to 3. Total scores rang from 0 (minimum) to 39 (maximum) for each drug the participant reports using.
(Frequency of) Events (i.e., Barriers) in Care Screening Questionnaire | Baseline
  Frequency of events that act as barriers to engagement in HIV care. Values: 9 items, range from 0 (not at all) to 2 (a great deal). Scoring: Higher scores = greater frequency of events that act as barriers to care engagement
Group-Based Medical Mistrust Scale | Throughout study completion: Baseline and 3-, 6- and 9-Month Follow-Up Post-Baseline
  Extent of mistrust in the medical system and healthcare providers, in general, based on the participant's and participant communities' beliefs and experiences.
  Values: 12 items, range from 12 (minimum) to 60 (maximum) Scoring: Greater scores = Greater levels of medical mistrust
Internalized AIDS-Related Stigma Scale | Throughout study completion: Baseline and 3-, 6-, and 9-Month Follow-Up Post-Baseline
  Extent to which the participant living with HIV holds negative beliefs about HIV and AIDS.
  Values: 6 items, range from 6 (minimum) to 30 (maximum). Scoring: Greater scores = greater degree of internalized stigma.
Cultural Assessment of Risk for Suicide (CARS) Minority Stress Subscale | Throughout study completion: Baseline and 3-, 6-, and 9-Month Follow-Up Post-Baseline
  Extent of minority stress, or forms of enacted stigma as stressors, experience by the participant.
  Values: 5 items in this subscale, range of 5 (minimum) to 30 (maximum). Scoring: Greater scores = greater minority stress; last item must be reverse coded.
Everyday Discrimination Scale | Baseline
  Extent of everyday discrimination, from the extreme to the mundane, experienced by the participant.
  Values: 9 items, range of 9 (minimum) to 54 (maximum). Scoring: Greater scores = more frequent perceived/experienced discrimination; has a follow-up question that allows participants to attribute experiences of discrimination to various aspects of identity.